CLINICAL TRIAL: NCT07098338
Title: An Open-Label, Multi-Drug, Multi-Centre, Phase II Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Antitumour Activity of Novel Combinations in Participants With Locally Advanced or Metastatic Non-Small Cell Lung Cancer (LIBRA)
Brief Title: A Study of Novel Combinations in Non-Small Cell Lung Cancer (NSCLC)
Acronym: LIBRA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D6187C00001
Record Dates: First submitted 2025-07-04; First posted 2025-08-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer(NSCLC); Antibody-Drug Conjugates (ADCs); T-cell immunoreceptor with Ig and Immunoreceptor Tyrosine-based Inhibition Motif (ITIM) domains (TIGIT); Programmed death-ligand 1 (PD-L1)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sub-study 1, investigate rilvegostomig± ramucirumab in 1L non-AGA NSCLC with PD-L1 ≥50% (Experimental): Participants will receive rilvegostomig ± ramucirumab until RECIST 1.1-defined radiological progression, unacceptable toxicity, withdrawal of consent, or other discontinuation criterion
  Interventions: Drug: Rilvegostomig; Drug: Ramucirumab
- Sub-study 2, investigate rilvegostomig + ramucirumab in 1L non-AGA NSCLC with PD-L1 1-49% (Experimental): Participants will receive rilvegostomig + ramucirumab until RECIST 1.1-defined radiological progression, unacceptable toxicity, withdrawal of consent, or other discontinuation criterion
  Interventions: Drug: Rilvegostomig; Drug: Ramucirumab
- Sub-study 3, investigate Dato-DXd + ramucirumab ± rilvegostomig in 2/3L AGA+ NSCLC (Experimental): Participants will receive Dato-DXd + ramucirumab ± rilvegostomig until RECIST 1.1-defined radiological progression, unacceptable toxicity, withdrawal of consent, or other discontinuation criterion
  Interventions: Drug: Rilvegostomig; Drug: Ramucirumab; Drug: Dato-DXd

INTERVENTIONS:
Drug: Rilvegostomig — Rilvegostomig will be administered as IV infusion.
  Other Names: AZD2936
Drug: Ramucirumab — Ramucirumab will be administered as IV infusion.
  Other Names: Cyramza
Drug: Dato-DXd — Dato-DXd will be administered as IV infusion.
  Other Names: DS-1062
  Arms: Sub-study 3, investigate Dato-DXd + ramucirumab ± rilvegostomig in 2/3L AGA+ NSCLC

SUMMARY:
This is a Phase II, multi-center, open-label platform study evaluating novel combination treatment options in participants with locally advanced or metastatic NSCLC. The study will consist of several sub-studies, each evaluating the safety, tolerability, and preliminary antitumour activity of various treatment combinations. This study will be conducted in approximately 80 centers globally across 10 countries.

DETAILED DESCRIPTION:
The master protocol will include 3 sub-studies, each focused on a specific disease population.

* Sub-study 1 will investigate rilvegostomig± ramucirumab in 1L non-actionable genomic alterations (AGA) NSCLC with PD-L1 ≥50%.
* Sub-study 2 will investigate rilvegostomig + ramucirumab in 1L non-actionable genomic alterations (AGA) NSCLC with PD-L1 1-49%.
* Sub-study 3 will investigate Dato-DXd + ramucirumab ± rilvegostomig in 2/3L AGA+

Each sub-study may include 2 parts (unless stated in the individual sub study protocols): Part A: one or more Safety Run-in cohort(s), and Part B: one or more Dose Expansion cohort(s).

ELIGIBILITY:
Inclusion Criteria for All Sub-studies:

* Participant must be ≥ 18 years of age at the time of signing the ICF
* WHO/ECOG performance status of 0 or 1
* At least 1 lesion that qualifies as a RECIST 1.1 Target Lesion (TL) at baseline.
* Adequate bone marrow and organ function
* Life expectancy ≥ 12 weeks
* Provision of acceptable tumour tissue

Specific Inclusion Criteria for Sub-Study 1 and Sub-Study 2:

* Histologically or cytologically documented advanced or metastatic NSCLC
* PD-L1 TC ≥ 1% (TC≥ 50% for sub-study 1, 1-49% for sub-study 2)
* Absence of sensitizing EGFR mutations or ALK rearrangements. No known other Actionable Genomic Alterations(AGAs)

Specific Inclusion Criteria for Sub-Study 3:

* Histologically or cytologically documented advanced or metastatic non-squamous NSCLC
* Documented positive AGA and had progressed on prior targeted therapy

Exclusion Criteria for All Sub-studies:

* As judged by the investigator, any severe or uncontrolled systemic diseases, in the investigator's opinion, makes it undesirable for the participant to participate in the study or that would jeopardise compliance with the protocol
* Active or prior documented autoimmune or inflammatory disorders
* Persistent toxicities (CTCAE Grade ≥ 2) (NCI CTCAE v5.0) caused by previous anti cancer therapy, excluding alopecia.
* Spinal cord compression or leptomeningeal carcinomatosis for sub-study 1 and sub-study 2. Unstable spinal cord compression for sub-study 3
* Unstable brain metastases
* History of another primary malignancy.
* Active infection, including TB and infections with HIV, HBV (verified by known positive HBsAg result), HCV.
* Uncontrolled or significant cardiac disease
* Receipt of prior systemic chemotherapy/chemoradiation/immunotherapy for advanced NSCLC for sub-study 1 and sub-study 2.
* Prior exposure to immune-mediated therapy
* History of uncontrolled hypertension, and active bleeding diseases, and high risks of bleeding and disorders of coagulation
* Any concurrent anti-cancer treatment.
* Receipt of live, attenuated vaccine within 30 days prior to the first dose of study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2029-04-06 (Estimated); Study Completion 2029-04-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AE) and serious adverse events (SAE) | Through study completion, an average of 3 years
  To assess the safety and tolerability
Objective response rate (ORR) | Through study completion, an average of 3 years
  ORR is defined as the proportion of participants who have a confirmed CR (complete response) or confirmed PR (partial response) per RECIST 1.1

SECONDARY OUTCOMES:
Best Overall Response(BOR) | Through study completion, an average of 3 years
  BOR is the best response a participant has had following randomisation/start of dosing, but prior to starting any subsequent cancer therapy and up to and including RECIST progression or the last evaluable assessment in the absence of RECIST progression
Change in Target Lesion Tumor Size | Through study completion, an average of 3 years
  The best percentage change from baseline in Target Lesion tumour size is the largest decrease (or smallest increase) from baseline for a participant, using RECIST 1.1 assessments
Progression free survival (PFS) | Through study completion, an average of 3 years
  PFS is defined as the time from the start of treatment until the date of objective disease progression or death (by any cause in the absence of progression) per RECIST 1.1.
Disease Control Rate(DCR) at 12 Weeks | From Day 1 pre-dose to 12 weeks
  DCR at 12 weeks is defined as the percentage of participants who have a best objective response of confirmed CR or PR or who have SD for at least 11 weeks after start of treatment (to allow for an early assessment within the assessment window).
Duration Of Response (DoR) | Through study completion, an average of 3 years
  The DoR is defined as the time from the date of first documented objective response (which is subsequently confirmed) until date of first documented disease progression or death (by any cause in the absence of disease progression).
Overall Survival(OS) | Through study completion, an average of 3 years
  OS is defined as the time from the start of treatment until death due to any cause.
Serum concentration | Through study completion, an average of 3 years
  To assess the serum concentration of the novel anti-cancer agents in combination.
Maximum plasma drug concentration (Cmax) | Through study completion, an average of 3 years
  To assess the Cmax of the novel anti-cancer agents in combination.
Immunogenicity of study interventions in participants receiving treatment | Through study completion, an average of 3 years
  Presence of Anti Drug Antibodies（ADAs) for study interventions in serum/plasma

CONTACTS AND LOCATIONS:
Locations (48):
- United States (6):
  - Research Site, Santa Monica, California
  - Research Site, Santa Rosa, California
  - Research Site, Atlanta, Georgia
  - Research Site, Baltimore, Maryland
  - Research Site, Houston, Texas
  - Research Site, Fairfax, Virginia
- Australia (2):
  - Research Site, Nedlands
  - Research Site, Woodville
- Research Site, Toronto, Ontario, Canada
- China (16):
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Deyang
  - Research Site, Dongguan
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Linyi
  - Research Site, Mianyang
  - Research Site, Nanchang
  - Research Site, Shantou
  - Research Site, Shenyang
  - Research Site, Wuhan
  - Research Site, Zhengzhou
  - Research Site, Zhuhai
- Japan (10):
  - Research Site, Bunkyō City
  - Research Site, Fukuyama-shi
  - Research Site, Kobe
  - Research Site, Kurume-shi
  - Research Site, Kyoto
  - Research Site, Osaka
  - Research Site, Sakaishi
  - Research Site, Shinjuku-ku
  - Research Site, Wakayama
  - Research Site, Yokohama
- Research Site, Singapore, Singapore
- South Korea (5):
  - Research Site, Cheongju-si
  - Research Site, Namdong-gu
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Suwon
- Taiwan (5):
  - Research Site, Liuying
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (2):
  - Research Site, Bangkok
  - Research Site, Banphaeo

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/